CLINICAL TRIAL: NCT04598087
Title: Multiphasic Prehabilitation in Patients Undergoing Surgery for Head and Neck Cancer
Brief Title: Prehabilitation and Recovery After Head and Neck Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA-CC-20-0013
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Surgery
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental): - Tailored exercise prescription involving aerobic and resistance training, supported by a clinical exercise physiologist.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — The multi-phasic prehabilitation intervention involves three phases: Phase 1: Before surgery (typically ~25 days); Phase 2: The in-hospital phase (typically 10-14 days); Phase 3: Discharge to 6-weeks after surgery.

SUMMARY:
Implementing a multiphasic, multimodal prehabilitation intervention for people undergoing surgery with free flap reconstruction for the treatment of head and neck cancer.

DETAILED DESCRIPTION:
BACKGROUND: Head and neck cancer (HNC) is the 7th most common cancer worldwide, and treatment often involves surgery. HNC surgery is intensive, complications are common, and quality of life (QOL) is negatively impacted. Support must be expanded to not only help patients survive HNC but to recover faster and live well following surgery. Prehabilitation, or optimizing a patient's condition before surgery, is a key opportunity to integrate supportive care early in the clinical care pathway for this underserved patient group. RESEARCH DESIGN AND METHODS: Using a mixed-methods approach, the aims of this hybrid implementation-effectiveness study are to (i) implement a multiphasic exercise prehabilitation program for HNC patients in a real-world setting and describe factors influencing implementation across the phases; (ii) determine the safety and tolerability of a multiphasic exercise prehabilitation program for HNC patients; (iii) explore the potential benefits of a multiphasic exercise prehabilitation program for HNC patients, and (iv) build a systematic screening and referral pathway into exercise oncology resources post-operatively. Outcomes are detailed below and include patient-reported outcomes, physical function, mobility (step count) and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Histologically verified primary head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, larynx, or in lymph nodes of the neck from an unknown primary tumour
* Scheduled to undergo oncologic resection or resection for benign disease with free flap reconstruction
* Approval received from a clinical exercise physiologist (CSEP-CEP) and/or clinician
* Ability to provide written informed consent and understand study information in English

Exclusion Criteria:

* Neurological or musculoskeletal co-morbidity inhibiting exercise
* Diagnosed psychotic, addictive, or major cognitive disorders
* Severe coronary artery disease (Canadian Cardiovascular Society class III or greater)
* Significant congestive heart failure (New York Heart Association class III or greater)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life: Functional Assessment of Cancer Therapy-Head and Neck Version 4 (FACT-H&N) | Baseline, 6 weeks, 6 months and 12 months after surgery (6 months is primary).
  Total score ranges from 0-156. A higher score is a better outcome.

SECONDARY OUTCOMES:
Weekly step counts | Phase 1 (before surgery)
  Total weekly step counts, measured using the Garmin vivosmart® 4
Weekly "intensity minutes" | Phase 1 (before surgery)
  Total weekly "intensity minutes", measured using the Garmin vivosmart® 4
Weekly step counts | Phase 3 (0-6 weeks after hospital discharge)
  Total weekly step counts. Garmin vivosmart® 4
Weekly "intensity minutes" | Phase 3 (0-6 weeks after hospital discharge)
  Total weekly step counts, measured using the Garmin vivosmart® 4
Self-reported moderate and strenuous physical activity score: Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Pre-intervention, 6 weeks after surgery, 6 and 12 months after cancer treatment
  [moderate frequency per week × 5] + [strenuous frequency per week × 9]. A higher score indicates more physical activity. The minimum score is 0, the maximum is dependent on the participant's frequency of physical activity.
Self-reported physical activity (leisure score index): Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline, 6 weeks after surgery, 6 and 12 months after cancer treatment
  [mild frequency per week × 3] + [moderate frequency per week × 5] + [strenuous frequency per week × 9]. A higher score indicates more physical activity. The minimum score is 0, the maximum is dependent on the participant's frequency of physical activity.
Fatigue severity: Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F). Total score. | Baseline, 10-14 days after surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Total score ranges from 0-52. Higher score means lower fatigue severity.
Anxiety score: Hospital Anxiety and Depression Scale (HADS) | Baseline, 10-14 days after surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Score ranges from 0-21, a higher score means more anxiety symptoms.
Depression score: Hospital Anxiety and Depression Scale (HADS) | Baseline, 10-14 days after surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Score ranges from 0-21, a higher score means more depressive symptoms.
Symptom burden: Edmonton Symptom Assessment System (ERAS-r). | Baseline, 10-14 days after surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Each item scored from 0 (no symptom) to 10 (worst possible symptom)
Self-reported health status: EQ VAS (visual analogue) score | Baseline, 10-14 days after surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Score ranges from 0 (worst health) to 100 (best health).
Single-leg balance (s) | Before surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Timed single-limb stance, both legs where tolerable, eyes open and closed where tolerable, up to a maximum of 45 seconds.
Lower-limb muscular endurance (number of sit-to-stands) | Before surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Thirty second sit-to-stand test
Functional exercise capacity (total steps) | Before surgery, 6 weeks after surgery, 6 and 12 months follow-up
  Two-minute step test
Hospital length of stay (total number of days) | The in-hospital period after surgery (from surgery to hospital discharge)
  Part of routine clinical data collection with the Calgary Head & Neck Enhanced Recovery Program.
Number of complications | Within 1 year after surgery.
  Part of routine clinical data collection with the Calgary Head & Neck Enhanced Recovery Program.
Mobilization after surgery (i) | The mean of the hospital period after surgery (typically 10-14 days)
  Mean daily step count. Garmin vivosmart® 4
Mobilization after surgery (ii) | The in hospital period after surgery (typically 10-14 days)
  Total daily step counts. Garmin vivosmart® 4

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Culos-Reed, PhD, Principal Investigator — nculosre@ucalgary.ca
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagoner CW, Daun JT, Danyluk J, Twomey R, Murphy L, Peterson M, Gentleman E, Capozzi LC, Francis GJ, Chandarana SP, Hart RD, Matthews TW, McKenzie D, Matthews J, Nakoneshny SC, Schrag C, Sauro KM, Dort JC, Manaloto V, Burnett L, Chisholm A, Lau H, Culos-Reed SN. Multiphasic exercise prehabilitation for patients undergoing surgery for head and neck cancer: a hybrid effectiveness-implementation study protocol. Support Care Cancer. 2023 Nov 28;31(12):726. doi: 10.1007/s00520-023-08164-w. PMID 38012345